CLINICAL TRIAL: NCT06927739
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of Orticumab in Participants With Prior Myocardial Infarction Who Have Elevated Coronary Inflammation Based on FAI Score Assessed by CCTA
Brief Title: Focused Orticumab Research for Treating Inflammation in Coronary Arteries
Acronym: FORTIFY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abcentra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORT-2024-02
Record Dates: First submitted 2025-03-25; First posted 2025-04-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Acute Coronary Syndromes; Coronary Arterial Disease (CAD); Inflammation; Heart Disease; Myocardial Infarct; Atherosclerotic Coronary Vascular Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Inflammation; Heart Diseases; Myocardial Infarction | interventions — MLDL1278A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orticumab High Dose (Active Comparator)
  Interventions: Drug: Orticumab
- Orticumab Low Dose (Active Comparator)
  Interventions: Drug: Orticumab
- Placebo High Dose (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo Low Dose (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orticumab — Orticumab treatment for 24 weeks for post MI population
  Other Names: MLDL1278a; BI204
  Arms: Orticumab High Dose; Orticumab Low Dose
Drug: Placebo — Placebo for 24 weeks for the post MI population
  Arms: Placebo High Dose; Placebo Low Dose

SUMMARY:
The goal of this clinical trial is to determine the clinical effect of orticumab treatment on inflammation in study participants with prior myocardial infarction who have elevated coronary inflammation based on CCTA. The main question it aims to answer is:

Clinical effects of orticumab treatment on inflammation of the coronary artery parameters measured with CCTA

Researchers will compare the effects with placebo group after 6 months of treatment

Participants will Keep the planned study visit appointments Provide complete information about medical and medical history Speak to the study doctor before changing any of non-study treatments, including starting new medications, receiving any vaccinations, or setting out to join any other clinical studies

DETAILED DESCRIPTION:
Participants will have the opportunity to participate in a Day 14 sub study. Participants who enroll in this optional sub study will have safety assessment (AE monitoring) and a blood sample obtained for serum orticumab concentration measurement, ADA titer, clinical safety labs and cardiometabolic and inflammation biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must provide informed consent before any study specific activities are performed, must be able and willing to meet all requirements for randomization and must adhere to the schedules of activities.
2. Participant must be >180 days after presumed type-1 myocardial infarction (i.e., due to plaque rupture or erosion, either STEMI or NSTEMI) without subsequent unstable or severe angina (Canadian Cardiovascular Society Class 3 or 4) at the time of enrollment. Participants who have undergone PCI are allowed.
3. Participant must be on a stable cardiovascular treatment regimen consistent with local treatment guidelines for post-AMI patients (such as maximally tolerated statin and/or PCSK9 inhibitor medication for LDL reduction, antiplatelet medication, and hypertension treatment).
4. Participant must have an evaluable, pre-randomization CCTA with one of the following:

   1. A quantifiable Fat Attenuation Index (FAI) Score greater than or equal to the 50th centile (per reference standard) for their age group in at least two coronary arteries or
   2. A quantifiable Fat Attenuation Index (FAI) Score greater than or equal to the 75th centile (per reference standard) for their age group in at least one coronary artery
5. Participant must have body mass index (BMI) ≤ 40 kg/m2.
6. Adult male and female participants ≥18 years of age at the Screening Visit:

For female participants, the participant must not be pregnant or lactating and must be one of the following:

1. Postmenopausal, defined as amenorrhea for ≥ 12 months following cessation of all exogenous hormonal treatments; follicle stimulating hormone levels may be obtained at the investigator's discretion to confirm the participant is postmenopausal.
2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy. Tubal ligation is not considered as irreversible surgical sterilization.
3. Females of childbearing potential must have a negative serum or urine pregnancy test prior to the start of study drug. In the case of positive urine pregnancy testing, a negative serum sample for pregnancy testing, to confirm that the participant is not pregnant, must be obtained prior to start of study. They must also agree to use an adequate method of contraception from Baseline through the End of the study or for 30 days after the last dose of study drug (whichever is longer), which include the following: sexual abstinence (if preferred and usual lifestyle of the participant), condom with spermicidal gel, diaphragm with spermicidal gel, coil (intrauterine device), surgical sterilization, vasectomy, oral contraceptive pill, depo progesterone injections, progesterone implant (i.e., Implanon®), NuvaRing®, Ortho Evra®.

For male participants - Nonsterile male participants with sexual partners of childbearing potential must agree to use an adequate method of contraception, including sexual abstinence (if preferred and usual lifestyle of the participant), from Baseline through the End of the study.

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. Percutaneous coronary intervention or invasive diagnostic coronary angiogram planned after screening. Eligible participants who have an invasive diagnostic coronary angiogram performed in the absence of undergoing a new PCI may continue screening after the diagnostic angiogram has been performed or may be rescreened.
3. History of or planned coronary artery bypass grafting.
4. Documented episode of post-MI pericarditis in the 3 months before enrollment.
5. Presence of unstable or uncontrolled angina. Canadian CV society (CCS) angina class > 2.
6. Ongoing New York Heart Association Class IV HF.
7. Poorly controlled type 1 or type 2 diabetes mellitus (hemoglobin A1c >8.0%).
8. Increased risk of bleeding:

   1. With history or presence of any bleeding disorder.
   2. Signs of ongoing bleeding at screening (e.g., identified macroscopic bleeding, low hemoglobin presumed to be caused by bleeding) or high risk for major bleeding in accordance with the Investigator's assessment (participants taking clinically indicated antiplatelet and antithrombotic agents are acceptable).
   3. Known severe liver disease (e.g., >5´ upper limit of normal elevations in ALT and/or AST and other evidence of grade 3 or higher criteria applies such as from the CTCAE 5.0 guidelines).
9. History or presence of any of the following:

   1. Ongoing infection or febrile illness.
   2. Ongoing persistent or permanent atrial fibrillation or flutter.
   3. Cancer within 5 years before randomization, with the exception of non-melanoma skin cancer.
   4. Alcohol or substance abuse within 6 months before randomization, as judged by the investigator.
   5. Known history of hypersensitivity reactions to other biologics, to human IgG preparations, or to any component of orticumab, or ongoing severe allergy as judged by the investigator.
   6. Active positive results on screening for serum hepatitis C core antibody.
   7. Clinically documented hepatitis B or HIV.
10. Any clinically important abnormalities in clinical chemistry, hematology, coagulation parameters, as judged by the investigator.
11. Blood pressure values at screening (taken as the average of triplicate measurements):

    1. Systolic blood pressure < 90 mmHg or > 180 mmHg.
    2. Diastolic blood pressure > 100 mmHg.
    3. One triplicate retest (repeat of all 3) will be allowed during the same visit, at which point if the retest result is no longer exclusionary, the participant may be randomized
    4. Participants who are excluded based on elevated blood pressure may be rescreened following adequate treatment.
12. Participants with any of the following contraindications to CCTA.

    1. eGFR < 40 mL/min/1.73 m2 by the Chronic Kidney Disease Epidemiology Collaboration equation, or end stage renal disease treated with kidney transplant or renal replacement therapy.
    2. Allergy to iodinated contrast.
    3. History of contrast-induced nephropathy.
    4. Contraindication to nitroglycerin.
    5. Rapid heart rate that is uncontrolled by medical therapy.
    6. Inability to hold breath for at least 6 seconds.
13. Use of any of the following in the 180 days before randomization: IL-17 inhibitor, TNF inhibitor, IL-6 inhibitor, IL-1β inhibitor, methotrexate, cyclosporine, apremilast, colchicine, systemic steroids (topical steroid use is allowed).
14. COVID-19 vaccine within 90 days of screening CCTA.
15. Participants with a confirmed positive COVID-19 test within 90 days of screening CCTA.
16. Receipt of any investigational device or therapy within 6 months or 5 half-lives before screening (whichever is longer).
17. Planned participation in an additional investigational study of an intervention or biologic before the end of the follow-up period. Participation in observational studies or studies without investigational drugs or devices is allowed.
18. Participants who have previously been exposed to orticumab.
19. Participants who are legally institutionalized.
20. An employee or close relative of an employee of the sponsor, the CRO, or the study site, regardless of the employee or close relative's role.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-02-08 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline of the mean Fat Attenuation Index (FAI) score for the 3 coronary arteries (RCA, LAD and LCX) for orticumab compared to placebo at 24 weeks | 24 weeks
  Analysis of the mean FAI score around the coronary arteries will be performed from baseline and 6-month Coronary Computed Tomography Angiography (CCTA) procedures.
  FAI-score is a standardized measurement of coronary inflammation for each coronary artery (adjusted for age, sex as well as technical, biological, and anatomical characteristics) to allow individualized interpretation of the degree of coronary inflammation. FAI-Score is given at a scale of 0-100 with arbitrary unit.
  A higher FAI-score indicates an increase coronary inflammation.

SECONDARY OUTCOMES:
Change from baseline for coronary artery inflammation | 24 weeks
  Change from baseline for Fat Attenuation Index (FAI) parameters for orticumab compared to placebo after 24 weeks of treatment assessed by Coronary Computed Tomography Angiography (CCTA)
Change from baseline for CaRi-Heart score for orticumab compared to placebo at 24 weeks of treatment | 24 weeks
  CaRi-Heart Risk score represents the individualized patient risk of a fatal cardiac event at 8 years which incorporates the FAI score values into a prognostic model that includes information about CCTA-derived plaque metrics and clinical cardiovascular risk factors (diabetes, smoking, hypertension, hyperlipidemia).

OTHER OUTCOMES:
Change in coronary artery plaque burden accessed by Coronary Computed Tomography Angiography (CCTA) at 24 weeks | 24 weeks
  Change in coronary artery plaque parameters for orticumab compared to placebo at 24 weeks of treatment assessed by CCTA
Change in radiotranscriptomic biomarkers of coronary inflammation as assessed by Coronary Computed Tomography Angiography (CCTA) | 24 weeks
  Change from baseline on radiotranscriptomic biomarkers of coronary inflammation (e.g. C19RS) as measured by CCTA compared to placebo to determine the effects of orticumab treatment on coronary inflammation
Number and percent of participants with treatment-emergent adverse events (TEAEs), and any serious adverse events | 24 weeks
Incident of abnormal vital signs | 24 weeks
  Vital signs (including blood pressure and pulse rate) are measured and recorded at every visit to assess the safety and tolerability of orticumab in study participants. Incidence of abnormal vital signs will be recorded.
Number of participants with abnormal laboratory tests results and abnormal physical exam findings | 24 weeks

CONTACTS AND LOCATIONS:
Locations (38):
- United States (7):
  - Abcentra Investigational Site, Los Angeles, California
  - Abcentra Investigational Site, Torrance, California
  - Abcentra Investigational Site, Boca Raton, Florida
  - Abcentra Investigational Site, Richmond, Indiana
  - Abcentra Investigational Site, Louisville, Kentucky
  - Abcentra Investigational Site, Baltimore, Maryland
  - Abcentra Investigational Site, Midland, Michigan
- Czechia (5):
  - Abcentra Investigational Site, Ostrava, Moravian-Silesian Region
  - Abcentra Investigational Site, Pilsen, Plzeň Region
  - Abcentra Investigational Site, Prague, Praha 2
  - Abcentra Investigational Site, Prague, Praha 4
  - Abcentra Investigational Site, Brno, South Moravian
- Hungary (3):
  - Abcentra Investigational Site, Pécs, Baranya
  - Abcentra Investigational Site, Budapest, Central Hungary
  - Abcentra Investigational Site, Nyíregyháza, Szabolcs-Szatmár-Bereg
- Italy (5):
  - Abcentra Investigational Site, Caserta, Campania
  - Abcentra Investigational Site, Ferrara, Ferrara
  - Abcentra Investigational Site, Brescia, Lombardy
  - Abcentra Investigational Site, Milan, Lombardy
  - Abcentra Investigational Site, Pavia, Lombardy
- Poland (3):
  - Abcentra Investigational Site, Krakow, Lesser Poland Voivodeship
  - Abcentra Investigational Site, Wroclaw, Lower Silesian Voivodeship
  - Abcentra Investigational Site, Warsaw, Masovian Voivodeship
- Romania (3):
  - Abcentra Investigational Site, Baia Mare, Maramureş
  - Abcentra Investigational Site, Târgu Mureş, Mureș County
  - Abcentra Investigational Site, Timișoara, Timiș County
- Spain (4):
  - Abcentra Investigational Site, Córdoba, Andalusia
  - Abcentra Investigational Site, Madrid, Madrid
  - Abcentra Investigational Site, El Palmar, Murcia
  - Abcentra Investigational Site, Seville, Sevilla
- Sweden (3):
  - Abcentra Investigational Site, Danderyd, Stockholm County
  - Abcentra Investigational Site, Solna, Stockholm County
  - Abcentra Investigational Site, Gothenburg, Västra Götaland County
- United Kingdom (5):
  - Abcentra Investigational Site, London, Greater London
  - Abcentra Investigational Site, Manchester, Greater Manchester
  - Abcentra Investigational Site, Oxford, Oxfordshire
  - Abcentra Investigational Site, Bath, Somerset
  - Abcentra Investigational Site, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: Yes